CLINICAL TRIAL: NCT07013786
Title: Correlation Between Motor Control Dysfunction and Radiographic Parameter in Non Specific Chronic Low Back Pain
Acronym: MCD-RP-NSCLBP
Status: Not yet recruiting | Type: Observational
Sponsor: Mohammad Abdelazeem Darwish Saad (Other)
Responsible Party: Sponsor-Investigator, Mohammad Abdelazeem Darwish Saad, Correlation between motor control dysfunction and radiographic parameter in non specific chronic low back pain, Cairo University
Organization: Cairo University (Other)
Other Study IDs: CUFPT-TRIAL001
Record Dates: First submitted 2025-05-30; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Chronic Non Specific Low Back Pain
Keywords: Lumbar motor control dysfunction; Lumbopelvic parameters; Radiographic alignment; Transverse abdominis; Multifidus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSCLBP Patients: Patients aged 20-40 years diagnosed with non-specific chronic low back pain (NSCLBP). Participants will undergo assessment of lumbar motor control using a pressure biofeedback unit in two positions (crock lying and prone). Additionally, radiographic imaging will be performed to measure lumbopelvic parameters, including pelvic incidence (PI), pelvic tilt (PT), sacral slope (SS), and lumbar lordotic angle (LLA), to analyze their correlation with motor control dysfunction.
  Interventions: Diagnostic Test: Pressure biofeedback assessment

INTERVENTIONS:
Diagnostic Test: Pressure biofeedback assessment — Participants will be assessed for lumbar motor control using a pressure biofeedback unit (PBU) during the Abdominal Draw-In Maneuver (ADIM) in both crock lying and prone positions. This is a non-invasive test to evaluate deep core muscle function (TrA and MF) in patients with NSCLBP. No therapeutic intervention will be administered.

SUMMARY:
This study aims to investigate the relationship between motor control dysfunction (MCD) and radiographic parameters in non-specific chronic low back pain (NSCLBP). Participants will undergo specific clinical motor control tests and lumbar spine X-rays to evaluate the alignment and coordination of spinal and pelvic structures. Understanding this relationship may help improve rehabilitation strategies and reduce pain in affected individuals.

DETAILED DESCRIPTION:
Non-specific chronic low back pain (NSCLBP) is a common musculoskeletal condition associated with impaired neuromuscular coordination and motor control dysfunction (MCD). This study seeks to determine the correlation between MCD and radiographic parameters including pelvic incidence (PI), pelvic tilt (PT), sacral slope (SS), and lumbar lordotic angle (LLA).

A total of 64 participants aged 20-40 with NSCLBP will be evaluated at the Faculty of Physical Therapy, Cairo University. Motor control will be assessed using a pressure biofeedback unit in two positions (crock lying and prone) via the Abdominal Draw-in Maneuver (ADIM). Radiographic measurements will be taken using lateral lumbar spine X-rays in standing posture.

The aim is to identify whether poor activation of deep stabilizing muscles (Transverse Abdominus and Multifidus) correlates with abnormal pelvic alignment and altered spinal curvature. Outcomes may support more effective personalized rehabilitation protocols targeting neuromuscular control to improve spine-pelvis function in NSCLBP patients.

Statistical analysis will include Pearson correlation to test for associations between motor control test performance and radiographic angle values.

ELIGIBILITY:
Inclusion Criteria:

* . Patients diagnosed with non-specific chronic low back pain (NSCLBP) for more than 3 months

  * Age between 20 and 40 years
  * Both males and females
  * Body mass index (BMI) between 18.5 and 29.9
  * No physical therapy or medical treatment during the last 3 months
  * Able and willing to provide informed consent

Exclusion Criteria:

* • Patients with specific causes of low back pain (e.g., disc herniation, fractures, tumors, infections)

  * History of spinal or lower limb surgery or injury
  * Radiculopathy or neurological disorders affecting motor control
  * Diagnosed spinal deformities (e.g., scoliosis, spondyloarthropathy, ankylosing spondylitis)
  * Contraindications to X-ray (e.g., pregnancy)
  * Patients currently undergoing physical therapy or medical intervention

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Both males and females with NSCLBP are eligible to participate based on biological sex.
Study Population: Patients aged 20-40 years diagnosed with non-specific chronic low back pain (NSCLBP), recruited from the outpatient physical therapy clinic of Cairo University. Participants will be screened based on clinical and radiographic criteria to ensure eligibility and safety.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Lumbar Lordotic Angle | At baseline (during initial assessment visit)
  Radiographic measurement of the lumbar lordotic angle (LLA) in degrees to assess sagittal spinal alignment in patients diagnosed with non-specific chronic low back pain.
Pelvic Incidence Angle | At baseline (during initial assessment visit)
  Measurement of Pelvic Incidence Angle in degrees obtained from lateral radiographic imaging in patients with non-specific chronic low back pain.
Pelvic Tilt Angle | At baseline (during initial assessment visit)
  Assessment of pelvic tilt angle in degrees as part of the evaluation of lumbopelvic alignment in patients with non-specific chronic low back pain.
Sacral Slope Angle | At baseline (during initial assessment visit)
  Evaluation of sacral slope angle in degrees based on standard radiographic imaging in patients with non-specific chronic low back pain.
Lumbar Motor Control Assessment via Pressure Biofeedback during ADIM | At baseline (during initial assessment visit)
  Evaluation of lumbar motor control using pressure biofeedback during the Abdominal Draw-In Maneuver (ADIM) from crook lying and prone position. Pressure changes in mmHg will be recorded to assess the ability to maintain abdominal contraction.

CONTACTS AND LOCATIONS:
Overall Officials: Enas Fawzy Youssef, Phd,MSc,PSc, Principal Investigator — Cairo university- Faculty of physical therapy; Nevien Ezzat Elliethy, Phd,MSc,PSc, Principal Investigator — Cairo university- faculty of medicine,department of radiology; Tasneem Ehab Mohammad, Phd,MSc,PSc, Principal Investigator — Cairo university- Faculty of physical therapy

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and institutional policy. The study is conducted as part of an academic thesis and is not intended for open data sharing.

REFERENCES:
- [Background] Saragiotto BT, Maher CG, Yamato TP, Costa LO, Menezes Costa LC, Ostelo RW, Macedo LG. Motor control exercise for chronic non-specific low-back pain. Cochrane Database Syst Rev. 2016 Jan 8;2016(1):CD012004. doi: 10.1002/14651858.CD012004. PMID 26742533